CLINICAL TRIAL: NCT00471874
Title: An Observational Study to Examine the Relationship Between Rheumatoid Arthritis Disease Severity and Health Related Utility
Brief Title: Study Evaluating Health Related Utility in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0881X1-4427
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine in Australia what effect rheumatoid arthritis has on quality of life, and also to determine the costs that are associated with having rheumatoid arthritis.

DETAILED DESCRIPTION:
At a routine visit to the clinic, patients will be asked to answer questions about their symptoms, have a routine examination by the doctor, fill out a questionnaire that will ask questions about them, about their arthritis, about how it affects their well being and quality of life, and about treatment and costs. The questionnaire will take them about 30 minutes to complete. A blood test may also be required.

This ends the patient's involvement with the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with clinically defined rheumatoid arthritis diagnosed for at least 3 months
* Age 18 years or older
* Ability to complete the study documents in English

Exclusion Criteria:

· Current participation in a blinded trial of an investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-04; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com
Locations (4):
- Australia (4):
  - Darlinghurst, New South Wales
  - Wollongong, New South Wales
  - Maroochydore, Queensland
  - Malvern, Victoria